CLINICAL TRIAL: NCT04854850
Title: An Open-Label Study of the Apollo Device for Fatigue in Systemic Sclerosis
Brief Title: Apollo Device for Fatigue in Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robyn T. Domsic, MD, MPH (Other)
Collaborators: Apollo Neuroscience (Unknown)
Responsible Party: Sponsor-Investigator, Robyn T. Domsic, MD, MPH, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100104
Record Dates: First submitted 2021-03-20; First posted 2021-04-22 (Actual); Results first posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Systemic Sclerosis; Fatigue; Raynaud Phenomenon
Keywords: Systemic Sclerosis; Fatigue; Raynaud; Pain
MeSH Terms: conditions — Scleroderma, Systemic; Fatigue; Raynaud Disease; Pain

STUDY DESIGN:
Intervention Model Description: Open-label clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Apollo (Experimental): Participants will all receive Apollo devices.
  Interventions: Device: Apollo

INTERVENTIONS:
Device: Apollo — The Apollo System offers a convenient novel non-invasive, non-habit-forming solution to improve performance and recovery under stress in children and adults by delivering gentle wave-like vibrations to the body that improve autonomic nervous system balance in real time (Siegle & Rabin et al., under review). The gentle vibrations delivered by the Apollo System are extremely low intensity in that they are typically just barely noticeable or perceptible by the user. Additionally, the range of frequencies and intensities of the Apollo System have been safely used in numerous commercial products without adverse events reported, including sexual vibrators and massagers. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy.
  Other Names: Apollo System; Tuned Vibrartory Stimulation

SUMMARY:
The purpose of this study is to learn about the effect of Apollo (a vibrating wearable about the side of an Apple Watch) on fatigue, Raynaud symptoms, depression, quality of life, and disease symptoms in patients with systemic sclerosis.

SSc patients frequently have fatigue as a characteristic feature of their disease and fatigue negatively impacts quality of life (Haythornthwaite 2003, Richards 2003, Suarez-Almazor 2007, Basta 2017). The prevalence of fatigue among SSc patients is 75%, with 61% ranking fatigue among their top three most distressing complaints. Fatigue is also associated with poor sleep quality, greater pain and depressive symptoms (Sandusky 2009). We hypothesize that treatment with Apollo over 1 month will improve fatigue. If successful, the Apollo technology will be the first treatment option for fatigue and Raynaud's in this population.

DETAILED DESCRIPTION:
This is a study of the commercially available Apollo Neuro Wellness Device, which is not currently a medical device.

The device offers a convenient novel non-invasive, non-habit-forming solution to improve performance and recovery under stress in children and adults by delivering gentle wave-like vibrations to the body that improve autonomic nervous system balance in real time (Siegle & Rabin et al., under review). Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy.

A total of 30-40 patients will be enrolled and followed for 1 month, with baseline data collected before using Apollo and follow-up data collected after using the device. This clinical trial is open-label, meaning that all participants will receive Apollos and no placebos will be used. All participants will be allowed to continue underlying immunosuppressive and Raynaud therapy at stable doses during the trial. Since this is a pilot study, future larger controlled trials will be necessary to clearly demonstrate drug effectiveness.

At study registration there was an oversight and we did not include the secondary outcome of number of weekly Raynaud attacks. Raynaud visual analog scale (VAS) was not a secondary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Men or women aged 18 years and older
3. Diagnosis of Systemic sclerosis, as defined by 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc.
4. Baseline T score of 45 on the PROMIS-Fatigue scale.
5. Steady daily doses and any immunosuppressive medication, vasodilators, antidepressants and anxiolytic use for 4 weeks prior to baseline.
6. Currently owns and operates an iOS or Android smart phone regularly
7. Ability to comply with the clinical visits schedule and the study-related procedures.
8. Subjects who have struggled with symptoms of SSc (specifically fatigue and Raynauds) who have not received adequate symptom relief from prior treatment attempts (treatment-resistant) will be prioritized.

Exclusion Criteria:

1. Medical and surgical history

   * Major surgery within 8 weeks prior to screening
   * Participants with an active malignancy.
   * End-stage renal disease with an estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m2 (MDRD formula) or on dialysis at the screening visit
   * Hepatic insufficiency as defined by the Child-Pugh criteria
   * Hospitalization for any reason within four weeks of the study baseline visit.
   * History of sympathectomy or stellate ganglion block
   * Significant interstitial lung disease with FVC ≤ 50% of predicted, or DLCO (uncorrected for hemoglobin) ≤ 40% of predicted
   * Pulmonary hypertension with change in medications in the preceding four weeks
   * Actively prescribed standing doses of beta-blockers.
   * Actively prescribed standing doses of sedatives, hypnotics, opioids, or benzodiazepines.
   * Active or unstable psychotic disorder requiring current prescriptions of standing doses of antipsychotic medications
   * Active suicidal/homicidal ideation or a suicide or homicide attempt in the past year.
2. Pregnant or breastfeeding women
3. Other • Any other condition or therapy that would make the participant unsuitable for this study and will not allow participation for the full planned study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn T Domsic, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haythornthwaite JA, Heinberg LJ, McGuire L. Psychologic factors in scleroderma. Rheum Dis Clin North Am. 2003 May;29(2):427-39. doi: 10.1016/s0889-857x(03)00020-6. PMID 12841303
- [Background] Richards HL, Herrick AL, Griffin K, Gwilliam PD, Loukes J, Fortune DG. Systemic sclerosis: patients' perceptions of their condition. Arthritis Rheum. 2003 Oct 15;49(5):689-96. doi: 10.1002/art.11385. PMID 14558055
- [Background] Suarez-Almazor ME, Kallen MA, Roundtree AK, Mayes M. Disease and symptom burden in systemic sclerosis: a patient perspective. J Rheumatol. 2007 Aug;34(8):1718-26. Epub 2007 Jul 1. PMID 17611983
- [Background] Basta F, Afeltra A, Margiotta DPE. Fatigue in systemic sclerosis: a systematic review. Clin Exp Rheumatol. 2018 Jul-Aug;36 Suppl 113(4):150-160. Epub 2017 Dec 15. PMID 29303706
- [Background] Sandusky SB, McGuire L, Smith MT, Wigley FM, Haythornthwaite JA. Fatigue: an overlooked determinant of physical function in scleroderma. Rheumatology (Oxford). 2009 Feb;48(2):165-9. doi: 10.1093/rheumatology/ken455. Epub 2008 Dec 23. PMID 19106163
- [Derived] Hammaker K, Hu H, Laffoon M, Freno LA, Lafyatis R, Park Y, Domsic RT. Association of the Apollo Wearable With Fatigue, Raynaud Phenomenon, and Quality of Life in Patients With Systemic Sclerosis: A Pilot Study. J Rheumatol. 2025 Feb 1;52(2):158-164. doi: 10.3899/jrheum.2024-0551. PMID 39617410

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the University of Pittsburgh Scleroderma clinic
Groups:
- Apollo (Open-label): Participants will all receive Apollo devices.
  Apollo: The Apollo System offers a convenient novel non-invasive, non-habit-forming solution to improve performance and recovery under stress in children and adults by delivering gentle wave-like vibrations to the body that improve autonomic nervous system balance in real time (Siegle & Rabin et al., under review). The gentle vibrations delivered by the Apollo System are extremely low intensity in that they are typically just barely noticeable or perceptible by the user. Additionally, the range of frequencies and intensities of the Apollo System have been safely used in numerous commercial products without adverse events reported, including sexual vibrators and massagers. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy.
Period: Overall Study
Arm/Group | Apollo (Open-label)
Started | 25 (1st subject was enrolled remotely in July 2020)
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Apollo: Participants will all receive Apollo devices. Apollo: The Apollo System offers a convenient novel non-invasive, non-habit-forming solution to improve performance and recovery under stress in children and adults by delivering gentle wave-like vibrations to the body that improve autonomic nervous system balance in real time (Siegle & Rabin et al., under review). The gentle vibrations delivered by the Apollo System are extremely low intensity in that they are typically just barely noticeable or perceptible by the user. Additionally, the range of frequencies and intensities of the Apollo System have been safely used in numerous commercial products without adverse events reported, including sexual vibrators and massagers. Apollo vibrations activate touch receptors in the skin and are perceived as safety signals by the brain resulting in decreased stress, improved recovery, focus, and energy.
Arm/Group | Apollo
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
Diffuse Skin Involvement [Count of Participants; unit: Participants] — Defined by skin thickening proximal to the elbow or knee per physical examination.
  Participants | 9
History of Digital Ulcers [Count of Participants; unit: Participants] — Population: One participant did not have exam history available.
  Participants
    number analyzed (Participants) | 24
    (all) | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in PROMIS® Item Bank v1.0 - Fatigue - Short Form 13a (FACIT-Fatigue) at 4 Weeks (End-of-Study) Compared to Baseline
Description: The FACIT-Fatigue is a patient reported outcome of fatigue symptoms, with a score range of 13-65. Low scores indicate low levels of fatigue and high scores indicate high levels of fatigue. A T-score of 50 indicates the population mean with a standard deviation of 10. A lower t-score indicates less fatigue. There are no clinically relevant thresholds.
Time Frame: Change in FACIT-Fatigue from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Apollo (Open-label)
Number analyzed (Participants) | 25
T-score
  Change from baseline at 4 weeks | -7.0 (1.6)
  Baseline | 62.5 (5.7)
Statistical Analysis 1: Comparison: Apollo (Open-label); Test type: Other; p < 0.001, t-test, 2 sided

2. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI/SHAQ) at 4 Weeks (End-of-Study) Compared to Baseline
Description: The HAQ-D1/SHAQ is a patient-reported outcome of functional ability. It is a continuous scale with a results range of 0-3, with 0 meaning no disability and 3 meaning very severe disability.
Time Frame: Change in HAQ-D1/SHAQ from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apollo (Open-label)
Number analyzed (Participants) | 25
score on a scale | 0.12 (0.05)

3. Secondary Outcome: Change in Total Weekly Raynaud Phenomenon Attacks
Description: This is a difference in frequency count of total RP attacks per week from baseline to week 4 (end-of-study).
Time Frame: Change in total weekly attacks from baseline to 4 weeks
Measure: Mean (Standard Deviation); unit: attacks
Arm/Group | Apollo (Open-label)
Number analyzed (Participants) | 25
attacks | -3.4 (1.1)

4. Secondary Outcome: Change in the Raynaud Condition Score (RCS) at 4 Weeks (End-of-study) From Baseline
Description: The Raynaud Consition Score is a patient-reported outcome of a single question regarding Raynaud severity. It is a visual analog scale with a results range of 0-100. A score of 0 is no symptoms, and 100 is severe symptoms. It is recommended by OMERACT for assessment of Raynaud phenomenon.
Time Frame: From baseline to 4-week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apollo (Open-label)
Number analyzed (Participants) | 25
units on a scale | -0.76 (0.40)

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Apollo
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04854850/Prot_SAP_000.pdf